CLINICAL TRIAL: NCT00515814
Title: A Prospective Open Pilot Study With Functional Placebo-control to Evaluate the Efficacy and Tolerability/Safety of a Subretinal Implant in Blind Patients in Accordance With ICH/GCP Guidelines
Brief Title: Retina Implant Pilot Trial to Evaluate Safety & Efficacy in Blind Patients Having Degenerated Photo-receptors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Implant AG (Industry)
Responsible Party: Eberhart Zrenner / Prof. MD, Centre for Ophthalmology, Institute for Ophthalmic Research, University of Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RI-PT-2005; Retina Implant Project
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Retinitis Pigmentosa
Keywords: Legal blindness; Retinopathy pigmentosa; Hereditary condition; Photo-receptor degeneration; Retina implant; Subretinal implant
MeSH Terms: conditions — Retinitis Pigmentosa; Blindness | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1, 2 (Experimental): During measurement/test periods, investigator sets implant into ON or OFF condition without subjects knowledge of when device is active.
  Interventions: Device: Retina implant is surgically placed into subretinal position

INTERVENTIONS:
Device: Retina implant is surgically placed into subretinal position — Subretinal implant is either in ON or in OFF condition during test periods, such as FrACT, BaLM, grating, orientation & mobility.
  Other Names: Retina Implant, subretinal implant, vision prosthesis,; medical device for restoration of vision

SUMMARY:
The outcome of this trial will reveal the possibilities of the retinal implant to improve the situation of patients with hereditary retinal blindness caused by degenerations of the outer retina. This pilot study will give important information on safety and efficacy of sub-retinal implants.

DETAILED DESCRIPTION:
Although the design of the chip with a possible resolution of up to 1500 image points has the potential of providing object recognition, the quality of the image transmitted in this first human application cannot be foreseen. On the other hand clinical experience teaches us that even bare light recognition improves mobility of patients because of the ability to localize bright light sources such as windows or lamps.

ELIGIBILITY:
Inclusion Criteria:

* Hereditary retinal degeneration of the outer retinal layers with the retinal vessels still being perfused and pigments of mild to moderate density
* Blindness (at least monocular) or visual functions not appropriate for navigation/orientation
* Period of appropriate visual functions > 12 years / lifetime
* Visual acuity ≥ 0,05 in earlier life
* Electrically Evoked Phosphenes provide evidence of inner-retinal function.
* willing and able to give written informed consent

Exclusion Criteria:

* Any other ophthalmologic disease with relevant effect upon visual function (e.g. glaucoma, optic neuropathy, trauma, diabetic retinopathy, retinal detachment)
* Systemic disease that might imply considerable risk with regard to the surgical intervention and anesthesia (e.g. cardiovascular diseases, severe metabolic diseases)
* Neurological and/or psychiatric diseases (e.g. M. Parkinson, epilepsy, depression )
* Retina detected as too thin (< 100 µm) to expect required rest-functionality as shown via Optical Coherence Tomography (OCT).
* Women who are pregnant or nursing, or women of childbearing potential who are not willing to use a medically acceptable means of birth control for the duration of the study, or women unwilling to perform a pregnancy test before entering the study
* Participation in another clinical trial within the past 30 days

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Visual Acuity / Light-perception / Object-orientation are significantly improved with implant-ON versus OFF as shown via FrACT / BaLM / grating test (i.e. EFFICACY) | within implantation period
Patient treatment shows acceptable results (i.e. SAFETY) | within implantation period

SECONDARY OUTCOMES:
Activities of Daily Living are significantly improved with implant-ON versus OFF, as shown via Tasks of Daily Living test / Orientation & Mobility test (i.e. EFFICACY) | within implantation period
Non-acceptable surgical complications will terminate clinical study (i.e. SAFETY) | within implantation period

CONTACTS AND LOCATIONS:
Overall Officials: Eberhart - Zrenner, Prof.Dr.med., Principal Investigator — University Eye Hospital Tuebingen, Germany
Locations (2):
- Germany (2):
  - Eye Hospital Dresden-Friedrichstadt, Dresden
  - University Eye Hospital Tuebingen, Tübingen

REFERENCES:
- [Derived] Stingl K, Bartz-Schmidt KU, Gekeler F, Kusnyerik A, Sachs H, Zrenner E. Functional outcome in subretinal electronic implants depends on foveal eccentricity. Invest Ophthalmol Vis Sci. 2013 Nov 19;54(12):7658-65. doi: 10.1167/iovs.13-12835. PMID 24150759
- [Derived] Kusnyerik A, Greppmaier U, Wilke R, Gekeler F, Wilhelm B, Sachs HG, Bartz-Schmidt KU, Klose U, Stingl K, Resch MD, Hekmat A, Bruckmann A, Karacs K, Nemeth J, Suveges I, Zrenner E. Positioning of electronic subretinal implants in blind retinitis pigmentosa patients through multimodal assessment of retinal structures. Invest Ophthalmol Vis Sci. 2012 Jun 20;53(7):3748-55. doi: 10.1167/iovs.11-9409. PMID 22562517
- [Derived] Wilke R, Gabel VP, Sachs H, Bartz Schmidt KU, Gekeler F, Besch D, Szurman P, Stett A, Wilhelm B, Peters T, Harscher A, Greppmaier U, Kibbel S, Benav H, Bruckmann A, Stingl K, Kusnyerik A, Zrenner E. Spatial resolution and perception of patterns mediated by a subretinal 16-electrode array in patients blinded by hereditary retinal dystrophies. Invest Ophthalmol Vis Sci. 2011 Jul 29;52(8):5995-6003. doi: 10.1167/iovs.10-6946. PMID 21693599
- See also: patient self-help, support and advocacy organization — http://www.pro-retina.de